CLINICAL TRIAL: NCT01779349
Title: Bladder Outlet Obstruction Observation Using Dynamic Urine Vibration "Holter" With Correlation to Pressure Flow Study and Uroflowmetry.
Brief Title: Bladder Outlet Obstruction Observation Using Dynamic Urine Vibration "Holter"
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: sensor calibration and other R&D activities
Sponsor: P. Square Medical Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PSM - 005
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Bladder Outlet Obstruction
Keywords: benign prostatic hyperplasia (BPH); acoustic vibration
MeSH Terms: conditions — Urinary Bladder Neck Obstruction; Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dynamic Urine Vibration "Holter" (Experimental): each subject will undergo intervention for the diagnosis of bladder outlet obstruction first using the Dynamic Urine Vibration "Holter" and then urodynamically by pressure flow study
  Interventions: Device: Dynamic Urine Vibration "Holter"

INTERVENTIONS:
Device: Dynamic Urine Vibration "Holter" — each subject will undergo intervention for the diagnosis of bladder outlet obstruction first using the Dynamic Urine Vibration "Holter" and then urodynamically by pressure flow study

SUMMARY:
Current gold standard of bladder outlet diagnosis is pressure flow study. This study is invasive time consuming and requires expensive and complex set-up. In this study the investigators plan to evaluate an alternative technology that presumably is able to diagnose bladder outlet obstruction using a Dynamic Urine Vibration "Holter" based on a Urine Flow Vibration Analysis technology. The acoustic vibration sensor is a small device that records the vibration due to urine flow. The patient attaches the sensor to the penis using a disposable sensor patch for the duration of approximately one minute during one urination. The analysis is performed off-line and the results are compared to the results of a standard pressure flow study and to the standard free flowmetry test. The innovative technology for the diagnosis of bladder outlet obstruction is noninvasive, rapid and does not involve complex setup.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of benign prostatic hyperplasia (BPH)
* has indication for urodynamic evaluation
* Males 18 years and older
* Capability of understanding and having signed the informed consent form after full discussion of the research, nature of the treatment, and its risks and benefits.

Exclusion Criteria:

Any condition which, in the investigator opinion, makes the patient unsuitable

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Holter to confirm or exclude of bladder outlet obstruction | One recording at the time of urodynamic testing. (approximatly one minute)

SECONDARY OUTCOMES:
Efficacy of Holter to supply the free flowmetry test curve & values. | One recording at the time of urodynamic testing. (approximatly one minute)

CONTACTS AND LOCATIONS:
Overall Officials: Haim Matzkin, Prof., Principal Investigator — Urology Department Director, Tel Aviv Sourasky Medical Center
Locations (2):
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv